CLINICAL TRIAL: NCT00278174
Title: A Phase II Trial of Interferon Alpha-1b (IFN Alpha-1b) in Patients With Metastatic Clear Cell Renal Carcinoma
Brief Title: Interferon Alfa (IFN-Alpha-1b) in Renal Cancer With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald M. Bukowski, Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE15804; P30CA043703 (NIH); CCF-7752 (Other: Cleveland Clinic IRB); CASE15804 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — interferon-alfa-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant interferon alpha-1b

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of tumor cells and slow the growth of kidney cancer.

PURPOSE: This phase II trial is studying how well interferon alfa works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with metastatic renal clear cell carcinoma treated with interferon alfa-1b.

Secondary

* Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive interferon alfa-1b subcutaneously daily. Treatment continues in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed predominantly renal clear cell carcinoma

  * Clinical evidence of OR biopsy-proven metastatic disease to a site or sites distant from the primary tumor
* Must have measurable disease, defined as ≥ 1 unidimensionally measurable lesion measured as ≥ 20 mm with conventional techniques OR as ≥ 10 mm with spiral CT scan
* Good- or intermediate-risk category as defined by having ≤ 2 of the following factors:

  * Time from initial diagnosis to treatment < 1 year
  * Karnofsky performance status < 80%
  * Hemoglobin < lower limit of normal
  * Corrected calcium > 10.0 mg/dL
  * Lactate dehydrogenase (LDH) > 1.5 times upper limit of normal (ULN)
* No major clinical ascites or pleural effusion
* No CNS metastases by neurologic exam and CT scan or MRI

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.5 g/dL
* Creatinine ≤ 1.5 mg/dL (2.0 mg/dL in post-nephrectomy patients)
* Calcium normal
* Total bilirubin ≤ 1.5 mg/dL
* AST ≤ 3.0 times normal
* Alkaline phosphatase ≤ 2.5 times normal (10 times ULN in presence of bone metastases)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and for the duration of study treatment
* No history of serious cardiac arrhythmia, congestive heart failure, angina pectoris, or other severe cardiovascular disease (i.e., New York Heart Association class III or IV)
* No known positivity for HIV or hepatitis B surface antigen
* No history of seizure disorders
* No local and/or systemic infections requiring antibiotics within 28 days prior to study entry
* No other malignancy except basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the uterine cervix, or any malignancy treated with curative intent and in complete remission for > 3 years

PRIOR CONCURRENT THERAPY:

* No prior organ allografts
* No prior interferon
* No prior cytokine-based therapy for metastatic disease
* Prior radiotherapy is allowed for the control of pain from skeletal lesions provided treatment was completed > 28 days prior to study entry and patient has recovered
* No major surgery requiring general anesthesia within 28 days prior to study entry
* No more than 2 prior therapies for metastatic disease
* No concurrent palliative radiotherapy
* No concurrent chemotherapy
* No concurrent hormonal therapy except for hormones administered for nondisease-related conditions (e.g., insulin for diabetes)
* No concurrent steroid use except ongoing replacement therapy with physiologic doses of corticosteroids

  * No concurrent dexamethasone or other steroidal anti-emetics or anti-inflammatories
* No other concurrent anticancer therapy
* No concurrent aspirin or barbiturates
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Bukowski, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States